CLINICAL TRIAL: NCT02288793
Title: Prepared for Focused Assessment With Sonography in Trauma Examination?
Brief Title: Focused Assessment With Sonography in Trauma
Acronym: FAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Other Study IDs: FAST/2014/01
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Trauma; Ultrasonography
Keywords: attitudes; knowledge; examination
MeSH Terms: conditions — Wounds and Injuries; Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Survey — Survey about Knowledge and Attitude About Focused Assessment With Sonography in Trauma

SUMMARY:
The study evaluates the knowledge and attitude about Focused Assessment with Sonography in Trauma examination among medical students and medical staff in Poland.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study

Exclusion Criteria:

* not meet the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical staff: medical doctors, nurses, paramedics Medical students: PhD students, medicine students, nursing and paramedics studies
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Results of the Medical Knowledge Tool (Questionnaire) | 2 weeks
  Percentage of healthcare workers and medical students with appropriate knowledge assessed by 10- items questionnaire about basic information about Focused Assessment With Sonography in Trauma. For each correct answer participant receive 1 point (0-1 point scale).

CONTACTS AND LOCATIONS:
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland